CLINICAL TRIAL: NCT04343898
Title: Study of the Treatment and Outcomes in Critically Ill Patients With COVID-19
Acronym: STOP-COVID
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Montefiore Medical Center (Other); Baylor College of Medicine (Other); Baylor Health Care System (Other); Beth Israel Deaconess Medical Center (Other); University of Colorado, Denver (Other); Cook County Hospital (Other); The Cooper Health System (Other); Duke University (Other); Georgetown University (Other); Hackensack mountainside hospital (Unknown); Hackensack Meridian Health (Other); Indiana University Health Methodist Hospital (Other); Johns Hopkins University (Other); Loma Linda University (Other); Mayo Clinic (Other); Medical College of Wisconsin (Other); Northwestern University (Other); Weill Medical College of Cornell University (Other); NYU Langone Health (Other); Ochsner Health System (Other); Oregon Health and Science University (Other); Renown Health (Other); Rush University Medical Center (Other); New Jersey Medical School (Other); Rutgers Robert Wood Johnson Medical School (Other); Stanford University (Other); Temple University (Other); Tufts Medical Center (Other); Tulane University (Other); University of California, Davis (Other); University of California, Los Angeles (Other); University of California, San Diego (Other); University of California, San Francisco (Other); University of North Carolina, Chapel Hill (Other); University Hospitals Cleveland Medical Center (Other); University Medical Center of Southern Nevada (Other); University of Alabama at Birmingham (Other); University of Chicago (Other); University of Florida (Other); University of Illinois at Chicago (Other); University of Kentucky (Other); University of Miami (Other); University of Michigan (Other); University of Oklahoma (Other); University of Pennsylvania (Other); University of Pittsburgh Medical Center (Other); University of Tennessee (Other); University of Washington (Other); University of Texas, Southwestern Medical Center at Dallas (Other); Yale University (Other)
Responsible Party: Principal Investigator, David Leaf, Assistant Professor of Medicine, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2007P000003
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observational

SUMMARY:
Multicenter observational/registry study of the clinical features and outcomes of critically ill patients with COVID-19.

DETAILED DESCRIPTION:
The goals of this project are to determine the independent risk factors for hospital mortality and acute organ injury, and to identify treatment strategies associated with improved survival. Additionally, we will assess outcomes according to differences in geographic and institutional parameters.

ELIGIBILITY:
Inclusion Criteria (each of the following):

1. Adults (aged ≥18 years)
2. Laboratory-confirmed diagnosis of COVID-19
3. Hospitalized in the ICU for illness related to COVID-19

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults admitted to an intensive care unit for illness related to COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 5154 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
28-Day Mortality | 28-days from the day of ICU admission

SECONDARY OUTCOMES:
60-Day Mortality | 60-days from the day of ICU admission
90-Day Mortality | 90-days from the day of ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: David E Leaf, MD, MMSc, Principal Investigator — Brigham and Women's Hospital; Shruti Gupta, MD, MPH, Study Director — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Gupta S, Hayek SS, Wang W, Chan L, Mathews KS, Melamed ML, Brenner SK, Leonberg-Yoo A, Schenck EJ, Radbel J, Reiser J, Bansal A, Srivastava A, Zhou Y, Sutherland A, Green A, Shehata AM, Goyal N, Vijayan A, Velez JCQ, Shaefi S, Parikh CR, Arunthamakun J, Athavale AM, Friedman AN, Short SAP, Kibbelaar ZA, Abu Omar S, Admon AJ, Donnelly JP, Gershengorn HB, Hernan MA, Semler MW, Leaf DE; STOP-COVID Investigators. Factors Associated With Death in Critically Ill Patients With Coronavirus Disease 2019 in the US. JAMA Intern Med. 2020 Nov 1;180(11):1436-1447. doi: 10.1001/jamainternmed.2020.3596. PMID 32667668
- [Result] Gupta S, Wang W, Hayek SS, Chan L, Mathews KS, Melamed ML, Brenner SK, Leonberg-Yoo A, Schenck EJ, Radbel J, Reiser J, Bansal A, Srivastava A, Zhou Y, Finkel D, Green A, Mallappallil M, Faugno AJ, Zhang J, Velez JCQ, Shaefi S, Parikh CR, Charytan DM, Athavale AM, Friedman AN, Redfern RE, Short SAP, Correa S, Pokharel KK, Admon AJ, Donnelly JP, Gershengorn HB, Douin DJ, Semler MW, Hernan MA, Leaf DE; STOP-COVID Investigators. Association Between Early Treatment With Tocilizumab and Mortality Among Critically Ill Patients With COVID-19. JAMA Intern Med. 2021 Jan 1;181(1):41-51. doi: 10.1001/jamainternmed.2020.6252. PMID 33080002
- [Result] Hayek SS, Brenner SK, Azam TU, Shadid HR, Anderson E, Berlin H, Pan M, Meloche C, Feroz R, O'Hayer P, Kaakati R, Bitar A, Padalia K, Perry D, Blakely P, Gupta S, Shaefi S, Srivastava A, Charytan DM, Bansal A, Mallappallil M, Melamed ML, Shehata AM, Sunderram J, Mathews KS, Sutherland AK, Nallamothu BK, Leaf DE; STOP-COVID Investigators. In-hospital cardiac arrest in critically ill patients with covid-19: multicenter cohort study. BMJ. 2020 Sep 30;371:m3513. doi: 10.1136/bmj.m3513. PMID 32998872
- [Result] Gupta S, Coca SG, Chan L, Melamed ML, Brenner SK, Hayek SS, Sutherland A, Puri S, Srivastava A, Leonberg-Yoo A, Shehata AM, Flythe JE, Rashidi A, Schenck EJ, Goyal N, Hedayati SS, Dy R, Bansal A, Athavale A, Nguyen HB, Vijayan A, Charytan DM, Schulze CE, Joo MJ, Friedman AN, Zhang J, Sosa MA, Judd E, Velez JCQ, Mallappallil M, Redfern RE, Bansal AD, Neyra JA, Liu KD, Renaghan AD, Christov M, Molnar MZ, Sharma S, Kamal O, Boateng JO, Short SAP, Admon AJ, Sise ME, Wang W, Parikh CR, Leaf DE; and the STOP-COVID Investigators. AKI Treated with Renal Replacement Therapy in Critically Ill Patients with COVID-19. J Am Soc Nephrol. 2021 Jan;32(1):161-176. doi: 10.1681/ASN.2020060897. Epub 2020 Oct 16. PMID 33067383
- [Result] Molnar MZ, Bhalla A, Azhar A, Tsujita M, Talwar M, Balaraman V, Sodhi A, Kadaria D, Eason JD, Hayek SS, Coca SG, Shaefi S, Neyra JA, Gupta S, Leaf DE, Kovesdy CP; STOP-COVID Investigators. Outcomes of critically ill solid organ transplant patients with COVID-19 in the United States. Am J Transplant. 2020 Nov;20(11):3061-3071. doi: 10.1111/ajt.16280. Epub 2020 Sep 15. PMID 32844546
- [Result] Leaf RK, Al-Samkari H, Brenner SK, Gupta S, Leaf DE. ABO phenotype and death in critically ill patients with COVID-19. Br J Haematol. 2020 Aug;190(4):e204-e208. doi: 10.1111/bjh.16984. Epub 2020 Jul 30. No abstract available. PMID 32609874
- [Result] Flythe JE, Assimon MM, Tugman MJ, Chang EH, Gupta S, Shah J, Sosa MA, Renaghan AD, Melamed ML, Wilson FP, Neyra JA, Rashidi A, Boyle SM, Anand S, Christov M, Thomas LF, Edmonston D, Leaf DE; STOP-COVID Investigators. Characteristics and Outcomes of Individuals With Pre-existing Kidney Disease and COVID-19 Admitted to Intensive Care Units in the United States. Am J Kidney Dis. 2021 Feb;77(2):190-203.e1. doi: 10.1053/j.ajkd.2020.09.003. Epub 2020 Sep 19. PMID 32961244
- [Result] Easter SR, Gupta S, Brenner SK, Leaf DE. Outcomes of Critically Ill Pregnant Women with COVID-19 in the United States. Am J Respir Crit Care Med. 2021 Jan 1;203(1):122-125. doi: 10.1164/rccm.202006-2182LE. No abstract available. PMID 33026829
- [Result] Al-Samkari H, Gupta S, Leaf RK, Wang W, Rosovsky RP, Brenner SK, Hayek SS, Berlin H, Kapoor R, Shaefi S, Melamed ML, Sutherland A, Radbel J, Green A, Garibaldi BT, Srivastava A, Leonberg-Yoo A, Shehata AM, Flythe JE, Rashidi A, Goyal N, Chan L, Mathews KS, Hedayati SS, Dy R, Toth-Manikowski SM, Zhang J, Mallappallil M, Redfern RE, Bansal AD, Short SAP, Vangel MG, Admon AJ, Semler MW, Bauer KA, Hernan MA, Leaf DE; STOP-COVID Investigators. Thrombosis, Bleeding, and the Observational Effect of Early Therapeutic Anticoagulation on Survival in Critically Ill Patients With COVID-19. Ann Intern Med. 2021 May;174(5):622-632. doi: 10.7326/M20-6739. Epub 2021 Jan 26. PMID 33493012
- [Result] Shaefi S, Brenner SK, Gupta S, O'Gara BP, Krajewski ML, Charytan DM, Chaudhry S, Mirza SH, Peev V, Anderson M, Bansal A, Hayek SS, Srivastava A, Mathews KS, Johns TS, Leonberg-Yoo A, Green A, Arunthamakun J, Wille KM, Shaukat T, Singh H, Admon AJ, Semler MW, Hernan MA, Mueller AL, Wang W, Leaf DE; STOP-COVID Investigators. Extracorporeal membrane oxygenation in patients with severe respiratory failure from COVID-19. Intensive Care Med. 2021 Feb;47(2):208-221. doi: 10.1007/s00134-020-06331-9. Epub 2021 Feb 2. PMID 33528595
- [Result] Short SAP, Gupta S, Brenner SK, Hayek SS, Srivastava A, Shaefi S, Singh H, Wu B, Bagchi A, Al-Samkari H, Dy R, Wilkinson K, Zakai NA, Leaf DE; STOP-COVID Investigators. d-dimer and Death in Critically Ill Patients With Coronavirus Disease 2019. Crit Care Med. 2021 May 1;49(5):e500-e511. doi: 10.1097/CCM.0000000000004917. PMID 33591017
- [Result] Mathews KS, Soh H, Shaefi S, Wang W, Bose S, Coca S, Gupta S, Hayek SS, Srivastava A, Brenner SK, Radbel J, Green A, Sutherland A, Leonberg-Yoo A, Shehata A, Schenck EJ, Short SAP, Hernan MA, Chan L, Leaf DE; STOP-COVID Investigators. Prone Positioning and Survival in Mechanically Ventilated Patients With Coronavirus Disease 2019-Related Respiratory Failure. Crit Care Med. 2021 Jul 1;49(7):1026-1037. doi: 10.1097/CCM.0000000000004938. PMID 33595960
- [Result] Douin DJ, Shaefi S, Brenner SK, Gupta S, Park I, Wright FL, Mathews KS, Chan L, Al-Samkari H, Orfanos S, Radbel J, Leaf DE. Tissue Plasminogen Activator in Critically Ill Adults with COVID-19. Ann Am Thorac Soc. 2021 Nov;18(11):1917-1921. doi: 10.1513/AnnalsATS.202102-127RL. No abstract available. PMID 33872546
- [Result] Churpek MM, Gupta S, Spicer AB, Parker WF, Fahrenbach J, Brenner SK, Leaf DE; STOP-COVID Investigators. Hospital-Level Variation in Death for Critically Ill Patients with COVID-19. Am J Respir Crit Care Med. 2021 Aug 15;204(403-411):403-11. doi: 10.1164/rccm.202012-4547OC. PMID 33891529
- [Result] Vasquez CR, Gupta S, Miano TA, Roche M, Hsu J, Yang W, Holena DN, Reilly JP, Schrauben SJ, Leaf DE, Shashaty MGS; STOP-COVID Investigators. Identification of Distinct Clinical Subphenotypes in Critically Ill Patients With COVID-19. Chest. 2021 Sep;160(3):929-943. doi: 10.1016/j.chest.2021.04.062. Epub 2021 May 6. PMID 33964301
- [Result] Friedman AN, Guirguis J, Kapoor R, Gupta S, Leaf DE, Timsina LR; STOP-COVID Investigators. Obesity, inflammatory and thrombotic markers, and major clinical outcomes in critically ill patients with COVID-19 in the US. Obesity (Silver Spring). 2021 Oct;29(10):1719-1730. doi: 10.1002/oby.23245. Epub 2021 Aug 6. PMID 34109768
- [Result] Jezmir JL, Bharadwaj M, Chaitoff A, Diephuis B, Crowley CP, Kishore SP, Goralnick E, Merriam LT, Milliken A, Rhee C, Sadovnikoff N, Shah SB, Gupta S, Leaf DE, Feldman WB, Kim EY; STOP-COVID Investigators. Performance of crisis standards of care guidelines in a cohort of critically ill COVID-19 patients in the United States. Cell Rep Med. 2021 Sep 21;2(9):100376. doi: 10.1016/j.xcrm.2021.100376. Epub 2021 Jul 28. PMID 34337554
- [Result] Churpek MM, Gupta S, Spicer AB, Hayek SS, Srivastava A, Chan L, Melamed ML, Brenner SK, Radbel J, Madhani-Lovely F, Bhatraju PK, Bansal A, Green A, Goyal N, Shaefi S, Parikh CR, Semler MW, Leaf DE; STOP-COVID Investigators. Machine Learning Prediction of Death in Critically Ill Patients With Coronavirus Disease 2019. Crit Care Explor. 2021 Aug 19;3(8):e0515. doi: 10.1097/CCE.0000000000000515. eCollection 2021 Aug. PMID 34476402
- [Result] Merriam LT, Bharadwaj M, Jezmir JL, Leaf DE, Kim EY. Protocol to assess performance of crisis standards of care guidelines for clinical triage. STAR Protoc. 2021 Dec 17;2(4):100943. doi: 10.1016/j.xpro.2021.100943. Epub 2021 Nov 10. PMID 34786562
- [Result] Hsu CM, Gupta S, Tighiouart H, Goyal N, Faugno AJ, Tariq A, Raichoudhury R, Sharma JH, Meyer L, Kshirsagar RK, Jose A, Leaf DE, Weiner DE; STOP-COVID Investigators. Kidney Recovery and Death in Critically Ill Patients With COVID-19-Associated Acute Kidney Injury Treated With Dialysis: The STOP-COVID Cohort Study. Am J Kidney Dis. 2022 Mar;79(3):404-416.e1. doi: 10.1053/j.ajkd.2021.11.004. Epub 2021 Dec 4. PMID 34871701
- [Result] Toth-Manikowski SM, Caldwell J, Joo M, Chen J, Meza N, Bruinius J, Gupta S, Hannan M, Kagalwalla M, Madrid S, Melamed ML, Pacheco E, Srivastava A, Viamontes C, Lash JP, Leaf DE, Ricardo AC; STOP-COVID Investigators. Sex-related differences in mortality, acute kidney injury, and respiratory failure among critically ill patients with COVID-19. Medicine (Baltimore). 2021 Dec 17;100(50):e28302. doi: 10.1097/MD.0000000000028302. PMID 34918709
- [Result] Keene AB, Admon AJ, Brenner SK, Gupta S, Lazarous D, Leaf DE, Gershengorn HB; STOP-COVID Investigators. Association of Surge Conditions with Mortality Among Critically Ill Patients with COVID-19. J Intensive Care Med. 2022 Apr;37(4):500-509. doi: 10.1177/08850666211067509. Epub 2021 Dec 23. PMID 34939474
- [Result] Ricardo AC, Chen J, Toth-Manikowski SM, Meza N, Joo M, Gupta S, Lazarous DG, Leaf DE, Lash JP; STOP-COVID Investigators. Hispanic ethnicity and mortality among critically ill patients with COVID-19. PLoS One. 2022 May 18;17(5):e0268022. doi: 10.1371/journal.pone.0268022. eCollection 2022. PMID 35584148
- [Result] Sunderraj A, Cho C, Cai X, Gupta S, Mehta R, Isakova T, Leaf DE, Srivastava A; STOP-COVID Investigators. Modulation of the Association Between Age and Death by Risk Factor Burden in Critically Ill Patients With COVID-19. Crit Care Explor. 2022 Aug 29;4(9):e0755. doi: 10.1097/CCE.0000000000000755. eCollection 2022 Sep. PMID 36050992
- [Result] Vasbinder A, Meloche C, Azam TU, Anderson E, Catalan T, Shadid H, Berlin H, Pan M, O'Hayer P, Padalia K, Blakely P, Khaleel I, Michaud E, Huang Y, Zhao L, Pop-Busui R, Gupta S, Eagle K, Leaf DE, Hayek SS; STOP-COVID Investigatorsdouble dagger. Relationship Between Preexisting Cardiovascular Disease and Death and Cardiovascular Outcomes in Critically Ill Patients With COVID-19. Circ Cardiovasc Qual Outcomes. 2022 Oct;15(10):e008942. doi: 10.1161/CIRCOUTCOMES.122.008942. Epub 2022 Oct 4. PMID 36193749
- [Result] Green A, Rachoin JS, Schorr C, Dellinger P, Casey JD, Park I, Gupta S, Baron RM, Shaefi S, Hunter K, Leaf DE; STOP-COVID Investigators. Timing of invasive mechanical ventilation and death in critically ill adults with COVID-19: A multicenter cohort study. PLoS One. 2023 Jun 28;18(6):e0285748. doi: 10.1371/journal.pone.0285748. eCollection 2023. PMID 37379286